CLINICAL TRIAL: NCT07129213
Title: Validity and Reliability of the Balance Outcome Measure for Elder Rehabilitation
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Ebru Akbuğa Koç, Assistant Professor, Yeditepe University
Other Study IDs: Ydtp
Record Dates: First submitted 2025-07-31; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2023-01

CONDITIONS: Elderly; Geriatric

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group: healthy group

SUMMARY:
The aim of this study is to investigate the validity and reliability of the Balance Outcomes Scale in elder rehabilitation.

DETAILED DESCRIPTION:
The balance assessment scale in geriatric rehabilitation has been specially developed for use in the rehabilitation of geriatric individuals in terms of its efficiency in terms of time and resources, its adequate reflection of standing balance structure, and its validity and sensitivity to change. The Balance Assessment Scale in Geriatric Rehabilitation consists of the Step Test, Timed Up and Go Test, Functional Reach Test, and Static Balance Test while standing with eyes closed. These measurements can be evaluated by physical therapists to assess the fundamental areas of standing balance structure (static, dynamic, functional). Subsequently, the performance in each of these four measurements is converted into a 5-point ranking scale from 0 to 4, with 4 representing good balance performance, resulting in a total score out of 16. This scale demonstrates high internal consistency (Cronbach's alpha = 0.87) and has good validity with the motor component of the Functional Independence Scale and the Modified Old Age Mobility Scale. However, its validity and reliability in Turkish have not yet been investigated. The aim of this study is to investigate the validity and reliability of the Balance Outcomes Scale in geriatric rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a Mini-Mental Evaluation Test result of 24 and above

Exclusion Criteria:

* amputated individuals or those who have a disease such as paraplegia or tetraplegia that have walking problems
* cannot receive the necessary commands for the study.

Ages: 60 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy group
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
step test | 3 months
timed up and go | 3 months
  timed up and go
functional reach test | 3 months
  functional reach test
timed static stance | 3 months
  timed static stance
berg balance scale | 3 months
  berg balance scale
Mini mental test | 3 months
  Mini mental test

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No